

### Statistical Analysis Plan

NCT Number: NCT03729609

Title: General Drug Use Surveillance Protocol General Drug Use Surveillance for ADCETRIS Intravenous Infusion 50 mg "Untreated CD30-Positive Hodgkin's

Lymphoma"

Study Number: C25018

Document Version and Date: version 1.0 / 26-Jan-2023 (Final Analysis), version 1.0 /

07-Sep-2023 (final analysis additional analysis)

Certain information within this document has been redacted (ie, specific content is masked irreversibly from view) to protect either personally identifiable information or company confidential information.

Note; This document was translated into English as the language on original version was Japanese.

### Statistical Analysis Plan

n a m e : Adcetris for Intravenous Infusion 50 mg Product

t i t l e : General use-results surveillance S t u d y

[Untreated CD30 positive Hodgkin's lymphoma]

: Takeda Pharmaceutical Company Limited.

ialuse only and subject to the applicable Terms of Use Proberty of Lan

version 1.0: January 26, 2023

| 1 | D & | | 2 |
|---|---|---|---|
| 1 | | ons of terms | 3 |
| | | t of Terms and Abbreviations | 3 |
| | | alysis Sets | 0, |
| | | mber of digits to be displayed | |
| | • | portant identified risks, important potential risks, and important missing information | 6 |
| 2 | | of medical institutions surveyed and the number and composition of patients | 2 |
| | enrolled | | 27 |
| | 2.1 Dis | position of patients characteristics ient characteristics nt | 7 |
| 3 | Patient of | characteristics | 9 |
| | 3.1 Pat | ient characteristics | 9 |
| 4 | Treatme | nt | .10 |
| | 4.1 Ad | ministration status of Adcetris D exposure | .10 |
| | 4.2 AV | D exposure | .10 |
| | 4.3 Ad | ministration status of G-CSF preparations | .10 |
| 5 | Safety a | nalysis | .12 |
| | J.1 OU. | rairence of adverse events, adverse arag readulens, and infections | • • • |
| | 5.1.1 | Incidence of adverse events | .12 |
| | | Occurrence Status of Adverse Reactions/Infections | |
| | 5.1.3 Adverse events, adverse reactions, and infections included in the safety | | |
| | | specifications | .13 |
| | 5.2 Occ | currence status of adverse events, adverse reactions, and infections in patients | |
| | | cluded from safety evaluation | .14 |
| | | Adverse events in patients excluded from safety evaluation | |
| | | Data on adverse reactions and infections in patients excluded from safety evaluation. | |
| | | iousness, CTCAE Grade (worst value), timing of onset, outcome, occurrence of | .10 |
| | • | verse events and adverse drug reactions/infections by causal relationship with deetris | 15 |
| | <i>5</i> .3.1 | Seriousness, CTCAE Grade (worst value), timing of onset, outcome, occurrence of | . 13 |
| | X-0.5.1 | adverse events by causal relationship with Adcetris | 15 |
| | 5.3.2 | Occurrence Status of Adverse Reactions/Infections by Seriousness, CTCAE Grade | .10 |
| | 3.3.2 | (Worst Value), Time of Onset, and Outcome | 16 |
| | 5.4 Occ | currence Status of Adverse Reactions/Infections by Patient Background and | |
| | | eatment Factors | 17 |
| | 5.4.1 | | . 1 / |
| | J. <del>4</del> .1 | and treatment details factor | 17 |

| 5.4.2 Occurrence Status of ADRs and Infections by Gender | 18 |
|---|---|
| 5.4.3 Occurrence Status of Adverse Reactions and Infections by Age Group | 19 |
| 5.4.4 Occurrence Status of Adverse Reactions/Infections by Presence/Absence of | 0 |
| Complication Renal Impairment | 19 |
| 5.4.5 Occurrence Status of Adverse Reactions/Infections by Presence/Absence of | 0) |
| Complication of Hepatic Impairment | 19 |
| 5.4.6 Occurrence Status of Adverse Reactions/Infections by Presence/Absence of Early | 19<br>19 |
| G-CSF Administration | .20 |
| 5.4.7 Occurrence Status of Adverse Reactions/Infections by Presence/Absence of Early | • |
| G-CSF Administration, Seriousness, CTCAE Grade (Worst Value), Time of Onset, | |
| and Outcome | 20 |
| 5.5 Administration status of Adcetris and AVD by outcome at the onset of adverse drug | |
| reactions/infections | 23 |
| 6 Efficacy analysis | 24 |
| 6.1 Antitumor response after the end of frontline therapy | 24 |
| 6.2 Antitumor effect after the end of frontline therapy by patient background factor and | |
| treatment factor | 24 |
| 7 Adverse reactions and infections in the additional pharmacovigilance plan | 26 |
| 7.1 Adverse reactions and infections included under the additional pharmacovigilance plan | |
| (Attached Form 12) | 26 |
| 8 Case summary in post-marketing surveillance | |
| 8.1 Case summary in post-marketing surveillance (Attached form 16) | |
| Preparation history (version control) | 28 |
| Property of Takeda: For non-comi | |
| <b>₹</b> 0′ | |
| Ž. | |
| Leo. | |
| the second secon | |
| DKO, | |

### **Definitions of terms**

### **List of Terms and Abbreviations**

- assessed by the investigator as having a causal relationship with Adcetris other than "Not related".

  In this statistical analysis plan, the term "adverse drug reactions/infections" will be used in the text or a serious adverse events.

  Serious adverse events.
- Serious adverse events: Adverse events assessed as "serious" by the investigator. Events listed in the MedDRA code list (PT code) using the Takeda Medically Significant AE List as the Important Medical Events List will be handled as serious events, even if the assessment by the investigator is "non-serious.
- Related to this product: An adverse event not related to Adcetris
- Not related to this product: Adverse events assessed as not related to Adcetris.
- Summary statistics: A general term for number of subjects, mean, standard deviation, maximum, minimum, and quartiles.
- Patients whose survey form was not collected: Patients whose survey form was not collected among registered patients.
- CRF collected patients: Patients whose CRF has been collected among registered patients.
- Days after treatment: Day-1 is defined as the day before the start of treatment with Adcetris, and Day 1 is defined as the day of the start of treatment with Adcetris.
- Duration of Adcetris treatment (days): End date of Adcetris treatment start date of Adcetris treatment +1
- Timing of onset of adverse events (or adverse drug reactions, etc.): Calculated as the date of onset of adverse events (or adverse drug reactions, etc.) – the start date of the first dose of Adcetris +1.
- Time from diagnosis of Hodgkin's lymphoma to first dose of Adcetris:
  - Actual number (unit: months) = (Year of the first administration of Adcetris Year of the diagnosis of Hodgkin's lymphoma) ×12+ (Month of the first administration of Adcetris – Month of the diagnosis of Hodgkin's lymphoma) If the month of the diagnosis is unknown, it should be calculated as January of the year described.

- Patients complicated with renal impairment: Patients for whom Takeda MedDRA query (Hereinafter referred to as TMQ) (Renal Disease) is entered in the disease name column.
- rems of Use Patients complicated with hepatic impairment: Patients with a complication corresponding to MedDRA standard query (hereinafter referred to as SMQ) code 20000005 (liver disorder SMQ [scope: narrow]) described in the disease name column.
- BMI(kg/m<sup>2</sup>): Calculated as weight (kg)/height (m)<sup>2</sup> (rounded off to the first decimal place).
- Treatment status
- Early treatment: G-CSF formulations administered within 5 days of the first dose of Adcetris.
  - Non-early administration: Administration of G-CSF on or after Day 6 of the first administration of Adcetris.
- Ation anistration anistration of the property of Takeda. For non-commercial use only and support of the property of Takeda. No early administration: Cases without administration of G-CSF preparations and cases with administration only other than early administration

### 1.2 **Analysis Sets**

The "safety evaluation population" and "efficacy evaluation population" will be set as the analysis

can be evaluated". Specifically, patients with locked CRFs who meet the following conditions will be excluded from the safety analysis set.

• Adcetris not administered
• Registration prior to the

- Enrollment after Day 31 of Adcetris treatment
- Unknown adverse event

aplan, "Patients evaluable as able for safety" is defined as active evaluation who meet the followation population.

a-target disease function or exclusion criteria violation

• Violation of exclusion criteria In this statistical analysis plan, "Patients evaluable for efficacy with no major protocol violations among patients evaluable for safety" is defined as "patients included in efficacy evaluation." Patients eligible for the safety evaluation who meet the following conditions will be excluded from the

### 1.3 Number of digits to be displayed

• Percentage (%)

Incidence of adverse events or adverse drug reactions:

Round the second decimal place and display to the second decimal place.

Other than the above:

Round the second decimal place and display to the first decimal place.

Summary statistics

Mean, 1st quantiles, median, 3rd quantiles:

The source data will be rounded to the first decimal place and displayed.

Standard deviation:

The data will be rounded to the second decimal place of the source data. Min, Max:

The same number of digits as that of the source data will be displayed.

### 1.4 Important identified risks, important potential risks, and important missing information

• Important identified risks

• Bone marrow depression: Events corresponding to MedDRA PT code 10029366 (neutrophil count decreased) or 10016288 (tebrile neutropenia). Among events corresponding to bone marrow depression, Grade ≥ 3 adverse events were collected in this study.

## Number of medical institutions surveyed and the number and composition of patients to the applicable Terms of Use that enrolled

### **Disposition of patients** 2.1

Survey for

General use-results survey

analysis:

Subjects for

All enrolled patients (patients enrolled)

analysis:

Analysis item:

Patients enrolled

Study sites

CRF not collected

Case report forms collected Patients excluded from safety

evaluation\*

Reason for exclusion (duplicate counting)

[Non-treatment with Adcetris, enrollment

before the contract period, enrollment after

the start date of treatment with Adcetris 31

days, unknown presence or absence of

adverse events, withdrawal of consent]

Safety analysis set

Patients excluded from efficacy

evaluation\*

Reason for exclusion [Off-label use, violation of inclusion criteria,

(duplicate counting) violation of exclusion criteria]

Efficacy analysis set

Method of

Property of Lakedai.

For the above analytical variables, the following analyses will be performed to

Analysis: prepare a case composition diagram.

> Also, the number of medical institutions surveyed will be shown for patients registered. A medical institution with a different department in the survey will be counted as 1 medical institution.

If there is no subject applicable to the reason for exclusion, 0 subject will be displayed.

For patients excluded from safety evaluation and patients excluded from efficacy evaluation, the number of patients by reason for exclusion will be tabulated and a list will be prepared.

\*"Patients excluded from safety evaluation" refer to patients excluded from" patients included in safety evaluation" among patients whose survey form was collected. Similarly, "patients excluded from efficacy evaluation" refers to

patients excluded from the "patients eligible for efficacy evaluation" among the

Property of Takeda: For non-commercial use only and subject to the applicable Tames of use

### 3 **Patient characteristics**

### **Patient characteristics** 3.1

Analysis Safety analysis population

population:

Sex Analysis item: [Male, female]

[Min <= - < 18, 18 <= - < 30, 30 <= -Age (years)

< 40, 40 <= - < 50, 50 <= - < 60, 60

- < 70, 70 <= - < 80, 80 <= - <= Max

[From the current month, the following Time from diagnosis of Hodgkin's lymphoma to first dose of Adcetris month, and the second and subsequent

months] (months)

[Lymph nodes, spleen, liver, lung, Lesion site (multiple counting)

bone, central nervous system, bone

marrow, skin, others]

Clinical Stage (Ann Arbor [Stage I, II, III, IV, unknown]

Classification)

BMI (kg/m<sup>2</sup>)

Presence or absence of B symptoms [Absent, present]

[0, 1, 2, 3, 4]**ECOG Performance Status** 

Treatment category (at the start of [Outpatient/inpatient]

treatment with Adcetris)

Complications [Absent, present]

Presence or absence of concomitant

renal impairment

Presence or absence of concomitant [Absent, present] hepatic impairment

Presence or absence of medical history [Absent, present, unknown]

 $Min \le -40.0, 40.0 \le -50.0,$ Body weight (kg)

 $50.0 \le -60.0, 60.0 \le -50.0,$ 

 $70.0 \le - \le Max$ , not measured

 $Min \le - < 18.5, 18.5 \le - < 25.0,$ 25.0 <= - < 30.0, 30.0 <= - <=

Max]

[Absent, present]

Pregnancy [Absent, present]

Breastfeeding (females only) [Absent, present]

For the above analytical variables, frequency tabulation of discrete data and

Property of Cakeda. Fo analysis: summary statistics of continuous data will be calculated.

### 4 Treatment

### 4.1 Administration status of Adcetris

Analysis Safety analysis population

population:

Analysis item : Adcetris initial dose (mg/kg)  $[Min \le -< 0.6, 0.6 \le -< 0.9, 0.9 \le -<$ 

- < 1.2, 1.2, 1.2 < - <= Max

Mean dose of Adcetris per  $[Min \le - < 0.6, 0.6 \le - < 0.9, 0.9 \le]$ 

administration (mg/kg) -<1.2, 1.2, 1.2<-<=Max

Adcetris dose per 2 weeks (mg/kg/2  $Min \le - < 0.6, 0.6 \le - < 0.9, 0.9 \le$ 

weeks) -<1.2, 1.2, 1.2 < -<= Max

Maximum number of doses [1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12]

Reasons for Discontinuation of [The treatment goal was achieved.,

Adcetris (Multiple Count) Onset of Grade ≥ 3 "neutropenia" or

"febrile neutropenia", The patient stopped visiting the hospital due to

transfer, pregnancy, Due to lack of

efficacy, Others

Method of For the above analytical variables, frequency tabulation of discrete data and

Analysis: summary statistics of continuous data will be calculated.

4.2 AVD exposure

Analysis Safety analysis population

population:

Analysis item: Initial dose of doxorubicin hydrochloride (mg/ m²)

Mean dose of doxorubicin hydrochloride per administration (mg/ m²)

Vinblastine sulfate initial dose (mg/ m<sup>2</sup>)

Mean dose of vinblastine sulfate per dose (mg/ m²)

Dacarbazine initial dose (mg/ m²)

Mean single dose of dacarbazine (mg/ m²)

Method of Summary statistics of continuous data will be calculated for the above analytical

Analysis: variables.

4.3 Administration status of G-CSF preparations

Analysis Safety analysis population

population:

Analysis item: Presence/absence of administration of [Absent, present]

G-CSF preparations

Property of Takeda: For non-commercial use only and subject to the applicable Temes of Use [With early administration, only Treatment status

11

### Safety analysis

### Occurrence of adverse events, adverse drug reactions, and infections

### 5.1.1 Incidence of adverse events

Analysis

population:

Analysis item:

To the above analytical variables, the following analyses should be performed.

(1) Number of patients with adverse events

(2) Number of adverse events

(3) I Analytical

method:

- (3) Incidence of adverse events
- (4) Type of adverse event

The method of accounting for each analysis is as follows.

[Number of patients with adverse events]

Number of patients with adverse events.

Number of adverse events

Number of adverse events experienced. If the same adverse event occurs more than once in the same patient, the total number of events will be tabulated.

[Incidence of adverse events]

Calculate as the number of patients with adverse events/the number of patients evaluable for safety ×100.

[Type of adverse event]

- Property of Lakedai. For non AEs will be coded using MedDRA/J. The data will be broadly classified by SOC and tabulated by PT. Note that cases in the SOC of "Investigations" will be summarized by HLGT (HLGT codes are sorted in ascending order, but not output) and by PT.
  - In the SOC, the number and percentage of patients with adverse events are presented in internationally agreed order of SOC. If the same SOC occurs more than once in the same subject, the subject will be counted as 1 subject in the SOC.
  - For PTs, the number of patients with adverse events and the incidence will be presented in ascending order of PT codes. If the same PT occurs more than once in the same patient, the patient will be counted as 1 patient for the PT.

### **5.1.2** Occurrence Status of Adverse Reactions/Infections

Safety analysis population Analysis

population:

Analysis item: Adverse reactions

, applicable Terms of Use Analytical For the above analytical variables, the following analyses should be performed.

method:

(1) Number of patients with adverse drug reactions

- (2) Number of adverse drug reactions
- (3) Incidence of adverse drug reactions
- (4) Types of adverse drug reactions, etc.

The method of accounting for each analysis is as follows.

[Number of patients with adverse drug reactions]

Number of patients with adverse drug reactions Number of adverse drug reactions

Number of adverse drug reactions. If the same adverse drug reaction, etc. occurs multiple times in the same patient, the total number of events will be tabulated.

### [Incidence of ADRs]

Calculate as the number of patients with adverse drug reactions/number of patients evaluable for safety ×100.

### Types of adverse reactions

- Adverse drug reactions will be coded using MedDRA/J. The data will be broadly classified by SOC and tabulated by PT. Note that cases in the SOC of "Investigations" will be summarized by HLGT (HLGT codes are sorted in ascending order, but not output) and by PT.
  - In the SOC, the number of patients with adverse drug reactions/infections and the incidence of them are described in internationally agreed order of SOC. If the same SOC occurs more than once in the same subject, the subject will be counted as 1 subject in the SOC.
- Property of Takedai. For non For PTs, the number of patients with adverse drug reactions/infections and the incidence of them will be described in ascending order of PT codes. If the same PT occurs more than once in the same patient, the patient will be counted as 1 patient for the PT.

### Adverse events, adverse reactions, and infections included in the safety specifications

### 5.1.3.1 Adverse events included in safety specifications

Analysis Safety analysis population population:

Analysis item: Adverse events included in safety specifications (important identified risks)

Stratification Seriousness [Serious, non-serious]

item:

Method of For the above analysis set, analyses should be performed in the same manner as

Analysis: in Section 5.1.1 for each of the subgroups of stratification factors by risk. If the

same SOC/PT occurs more than once in the same patient, the patient will be counted as 1 patient in the SOC/PT. However, if the seriousness is different, C case shall be counted for each of serious and non-serious cases. The risks covered should also follow the definition provided in the important identified

risks.

### 5.1.3.2 Incident Status of Adverse Reactions/Infections Included in Safety Specifications

Analysis Safety analysis population

population:

Analysis item: Adverse reactions corresponding to safety specifications (important identified

risks)

Stratification Seriousness [Serious, non-serious]

item:

Method of For the above analysis set, analyses should be performed in the same manner as

Analysis: in Section 5.1.2 for each of the subgroups of stratification factors by risk. If the

same SOC/PT occurs more than once in the same patient, the patient will be counted as 1 patient in the SOC/PT. However, if the seriousness is different, 1 case shall be counted for each of serious and non-serious cases. The risks covered should also follow the definition provided in the important identified

risks.

## 5.2 Occurrence status of adverse events, adverse reactions, and infections in patients excluded from safety evaluation

### 2.1 Adverse events in patients excluded from safety evaluation

Subjects Subjects excluded from safety evaluation

analyzed:

Analysis item: Adverse events

Method of For the above analytical variable, analyses should be performed in the same

Analysis: manner as in Section 5.1.1.

### 5.2.2 Data on adverse reactions and infections in patients excluded from safety evaluation

Subjects Subjects excluded from safety evaluation

analyzed:

Analysis item: Adverse reactions

Method of For the above analytical variable, analyses should be performed in the same

Analysis: manner as in Section 5.1.2.

### Seriousness, CTCAE Grade (worst value), timing of onset, outcome, occurrence of 5.3 adverse events and adverse drug reactions/infections by causal relationship with Adcetris

### 5.3.1 Seriousness, CTCAE Grade (worst value), timing of onset, outcome, occurrence of adverse events by causal relationship with Adcetris

Analysis Safety analysis population

population:

Analysis item: Adverse events

Stratification

Total

item:

Serious, non-serious] Seriousness

[Grade3, Grade4, Grade5] CTCAE Grade(worst)

[1 <= - <= 14, 15 <= - <= 28, 29 <= - <= Time of onset (days)

 $56, 57 \le -12, 113 \le -12 \le Max$ 

Time of onset (number of doses) [After the first dose to before the second

> dose, after the second dose to before the third dose, after the third dose to before the fifth dose, after the fifth dose to

before the ninth dose, and after the

ninth dose

Recovered/resolved,

recovering/resolving, not recovered/not

resolved, recovered/resolved with sequelae, death (due to the event),

unknown]

[Related, not related] Relationship to Adcetris

For the above analysis sets, analyses should be performed in the same manner as

in Section 5.1.1 for each of the subgroups of the stratification factors. If the

same SOC/PT occurs more than once in the same patient, the patient will be counted as 1 patient in the SOC/PT. However, for the same SOC, one case will

be adopted in the following order of priority, and the same PT will be adopted as

one case for the content of any of the stratification items in the following order of priority.

Seriousness: serious → non-serious

CTCAE Grade (worst): Grade5→Grade4→Grade3

Time of onset (days): 1 to 14 days  $\rightarrow$ 15 to 28 days  $\rightarrow$ 29 to 56 days  $\rightarrow$ 57 to

112 days  $\rightarrow \ge 113$  days

Time of onset (number of doses): After the first dose to before the second dose

→ After the second dose to before the third dose → After the third dose to before the fifth dose → After the fifth dose to before the ninth dose

the ninth dose and thereafter

Outcome: death (due to the event) → recovered with sequelae

recovered → recovering → recovered → unknown

Causal relationship with Adcetris: Related → Not related

## 5.3.2 Occurrence Status of Adverse Reactions/Infections by Seriousness, CTCAE Grade Use Only and (Worst Value), Time of Onset, and Outcome

Analysis Safety analysis population

population:

Analysis item: Adverse reactions

Stratification Total

item:

Time of onset (number of doses) Seriousness [Serious, non-serious]

[Grade3, Grade4, Grade5]

[1 <= - <= 14, 15 <= - <= 28, 29 <= - <=

56, 57 <= - <= 112, 113 <= - <= Max

[After the first dose to before the second dose, after the second dose to before the third dose, after the third dose to before

the fifth dose, after the fifth dose to

before the ninth dose, and after the

ninth dose]

[Recovered/resolved,

recovering/resolving, not recovered/not

resolved, recovered/resolved with sequelae, death (due to the event),

unknown]

Method of For the above analysis sets, analyses should be performed in the same manner as Analysis:

in Section 5.1.2 for each of the subgroups of the stratification factors. If the same SOC/PT occurs more than once in the same patient, the patient will be counted as 1 patient in the SOC/PT. However, for the same SOC, one case will be adopted in the following order of priority, and the same PT will be adopted as one case for the content of any of the stratification items in the following order of priority.

Seriousness: serious → non-serious

CTCAE Grade (worst value) : Grade5→Grade4→Grade3

Time of onset (days): 1 to 14 days  $\rightarrow$ 15 to 28 days  $\rightarrow$ 29 to 56 days

112 days  $\rightarrow \ge 113$  days

Timing of onset (number of doses): After the first dose to before the second dose  $\rightarrow$  After the second dose to before the third dose  $\rightarrow$  After the third dose to before the fifth dose → After the fifth dose to before the ninth dose → After the ninth dose and thereafter

Outcome: death (due to the event)  $\rightarrow$  recovered with sequelae  $\rightarrow$  not recovered → recovering → recovered → unknown

### Occurrence Status of Adverse Reactions/Infections by Patient Background and 5.4 **Treatment Factors**

### 5.4.1 Occurrence status of adverse drug reactions/infections by patient background factor and treatment details factor

Safety analysis population Analysis

population:

Analysis item: Adverse reactions

Stratification [Male, female] Property of Lakeda. For

 $Min \le - < 18, 18 \le - < 30, 30 \le -$ 

< 40, 40 <= - < 50, 50 <= - < 60, 60

<= - < 70, 70 <= - < 80, 80 <= - <=

Max

Time from diagnosis of Hodgkin's [From the current month, the following lymphoma to first dose of Adcetris month, and the second and subsequent

(months) months]

Lesion site (multiple counting) [Lymph nodes, spleen, liver, lung,

bone, central nervous system, bone

marrow, skin, others]

Clinical Stage (Ann Arbor [Stage I, II, III, IV, unknown] Classification)

Presence or absence of B symptoms [Absent, present] [0, 1, 2, 3, 4]**ECOG Performance Status** 

Treatment classification (at the start of

treatment with Adcetris)

[Outpatient/inpatient]

Presence or absence of complications [Absent, present]

Presence or absence of concomitant

renal impairment

[Absent, present]

Presence or absence of concomitant

hepatic impairment

[Absent, present]

cable Terms of Use [Absent, present, unknown] Presence or absence of medical history

Weight (kg)

BMI 
$$(kg/m^2)$$
 [Min  $\leq$  - < 18.5, 18.5  $\leq$  - < 25.0,

$$25.0 \le - < 30.0, 30.0 \le - \le Max$$

Adcetris initial dose (mg/kg)

$$\int [Min \le - < 0.6, 0.6 \le - < 0.9, 0.9]$$

$$<= - < 1.2, 1.2, 1.2 < - <= Max$$

 $[Min \le - < 0.6, 0.6 \le - < 0.9, 0.9]$ Mean Adcetris

administration (mg/kg) <= - < 1.2, 1.2, 1.2 < - <= Max

 $Min \le - < 0.6, 0.6 \le - < 0.9, 0.9$ Adcetris weeks

<= - < 1.2, 1.2, 1.2 < - <= Max(mg/kg/2weeks)

G-CSF Early administration [Absent, present]

Method of Analysis:

For the above analytical variable, the following analyses should be performed for each of the subgroups of the stratification factors.

Number of patients with adverse drug reactions

Incidence of adverse drug reactions

patients evaluable for safety ×100.

The method of accounting for each analysis is as follows.

[Number of patients with adverse drug reactions]

Number of patients with adverse drug reactions [Incidence of ADRs]

Calculate as the number of patients with adverse drug reactions/number of

## Property of Takeda. 5.4.2 Occurrence Status of ADRs and Infections by Gender

Safety analysis population Analysis

population:

Analysis item: Adverse reactions

Stratification Sex [Male, female]

item:

Method of For the above analysis sets, analyses should be performed in the same manner as

Analysis: in Section 5.1.2 for each of the subgroups of the stratification factors.

### 5.4.3 Occurrence Status of Adverse Reactions and Infections by Age Group

Analysis Safety analysis population

population:

Analysis item: Adverse reactions

Stratification Age (years)  $[Min \le - < 18, 18 \le - < 30, 30]$ 

item : <= -<40, 40 <= -<50, 50 <= -

< 60, 60 <= - < 70, 70 <= - < 80,

80 <= - <= Max

Method of For the above analysis sets, analyses should be performed in the same manner as

Analysis: in Section 5.1.2 for each of the subgroups of the stratification factors.

## 5.4.4 Occurrence Status of Adverse Reactions/Infections by Presence/Absence of Complication Renal Impairment

Analysis Safety analysis population

population:

Analysis item: Adverse reactions

Stratification Presence or absence of concomitant renal

[Absent, present]

item: impairment

Method of For the above analysis sets, analyses should be performed in the same manner as

Analysis: in Section 5.1.2 for each of the subgroups of the stratification factors.

### 5.4.5 Occurrence Status of Adverse Reactions/Infections by Presence/Absence of

Complication of Hepatic Impairment

Analysis Safety analysis population

population:

Analysis item: Adverse reactions

Stratification Presence or absence of concomitant

[Absent, present]

item: hepatic impairment

Method of For the above analysis sets, analyses should be performed in the same manner as

Analysis: in Section 5.1.2 for each of the subgroups of the stratification factors.

## 5.4.6 Occurrence Status of Adverse Reactions/Infections by Presence/Absence of Early G-CSF Administration

Analysis Safety analysis population

population:

Analysis item: Adverse reactions

Stratification Presence or absence of early G-CSF

item: administration

Method of For the above analysis sets, analyses should be performed in the same manner as

[Absent, present]

Analysis: in Section 5.1.2 for each of the subgroups of the stratification factors.

## 5.4.7 Occurrence Status of Adverse Reactions/Infections by Presence/Absence of Early G-CSF Administration, Seriousness, CTCAE Grade (Worst Value), Time of Onset, and Outcome

## 5.4.7.1 Occurrence Status of Adverse Reactions/Infections by Presence/Absence of Early G-CSF Administration and by Seriousness

Analysis Safety analysis population

population:

Analysis item: Adverse reactions

Stratification item Presence/absence of early G-CSF [Absent, present]

1: administration

Stratification item Seriousness [Serious, non-serious]

2:

Method of For the above analysis sets, the same analyses as those in Section 5.1.2 will be

analysis: performed for each stratum of Stratification Item 2 after stratifying for

Stratification Item 1. If the same SOC/PT occurs more than once in the same patient, the patient will be counted as 1 patient in the SOC/PT. However, for the same SOC, one case will be adopted in the following order of priority, and for the same PT, one case will be adopted for the content of any of the stratification

items 2 in the following order of priority.
Seriousness: serious → non-serious

## 5.4.7.2 Occurrence Status of Adverse Reactions/Infections by Presence/Absence of Early G-CSF Administration and CTCAE Grade (Worst)

Analysis Safety analysis population

population:

Analysis item: Adverse reactions

Stratification item Presence/absence of early G-CSF [Absent, present]

1: administration

Stratification item CTCAE Grade (worst) [Grade3, Grade4, Grade5]

2:

Method of For the above analysis sets, analyses should be performed in the same manner as

Analysis: in Section 5.4.7.1. If the same SOC/PT occurs more than once in the same

patient, the patient will be counted as 1 patient in the SOC/PT.However, for the same SOC, one case will be adopted in the following order of priority, and for the same PT, one case will be adopted for the content of any of the stratification

items 2 in the following order of priority.

CTCAE Grade (worst) : Grade5→Grade4→Grade3

## 5.4.7.3 Occurrence Status of Adverse Reactions/Infections by Presence/Absence of Early G-CSF Administration and Onset Time (Day)

Analysis Safety analysis population

population:

Analysis item: Adverse reactions

Stratification item Presence/absence of early G-CSF [Absent, present]

1: administration

Stratification item Time of onset (days)  $[1 \le - \le 14, 15 \le - \le 28, 29]$ 

2:

<= - <= Max \rightarrow

Method of For the above analysis sets, analyses should be performed in the same manner as

Analysis: in Section 5.4.7.1. If the same SOC/PT occurs more than once in the same

patient, the patient will be counted as 1 patient in the SOC/PT.However, for the same SOC, one case will be adopted in the following order of priority, and for the same PT, one case will be adopted for the content of any of the stratification

items 2 in the following order of priority.

Time of onset (days): 1 to 14 days  $\rightarrow$ 15 to 28 days  $\rightarrow$ 29 to 56 days  $\rightarrow$ 57 to

112 days  $\rightarrow \ge 113$  days

## 5.4.7.4 Occurrence Status of Adverse Reactions/Infections by Presence/Absence of Early G-CSF Administration and Onset Time (Dose)

Analysis Safety analysis population

population:

Analysis item: Adverse reactions

Stratification item Presence/absence of early G-CSF [Absent, present]

1: administration

Stratification item Time of onset (number of doses) [After the first dose to before the

2: second dose, after the second

dose to before the third dose, after the third dose to before the

fifth dose, after the fifth dose to

before the ninth dose, and after the ninth dose]

Method of For the above analysis sets, analyses should be performed in the same manner as

Analysis: in Section 5.4.7.1. If the same SOC/PT occurs more than once in the same

patient, the patient will be counted as 1 patient in the SOC/PT. However, for the same SOC, one case will be adopted in the following order of priority, and for the same PT, one case will be adopted for the content of any of the stratification items 2 in the following order of priority. Timing of onset (number of doses): After the first dose to before the second dose  $\rightarrow$  After the second dose to before the third dose  $\rightarrow$  After

the fifth dose to before the ninth dose - After the ninth dose and thereafter

5.4.7.5 Occurrence Status of Adverse Reactions/Infections by Presence/Absence of Early G-CSF Administration and Outcome

Analysis Safety analysis population

population:

Analysis item: Adverse reactions

Stratification item Presence/absence of early G-CSF [Absent, present]

1: administration

Stratification item Outcome [Recovered/resolved,

2: recovering/resolving, not

recovered/not resolved, recovered/resolved with sequelae, death (due to the

event), unknown]

Method of For the above analysis sets, analyses should be performed in the same manner as

Analysis: in Section 5.4.7.1. If the same SOC/PT occurs more than once in the same

patient, the patient will be counted as 1 patient in the SOC/PT.However, for the same SOC, one case will be adopted in the following order of priority, and for the same PT, one case will be adopted for the content of any of the stratification

items 2 in the following order of priority.

Outcome: death (due to the event)  $\rightarrow$  recovered with sequelae  $\rightarrow$  not

recovered  $\rightarrow$  recovering  $\rightarrow$  recovered  $\rightarrow$  unknown

## Plicable Leiths of Use Administration status of Adcetris and AVD by outcome at the onset of adverse drug 5.5 reactions/infections

Analysis Safety analysis population

population:

Analysis item: Adverse reactions

Stratification Presence or absence of change due to

item 1: this event

> [Dose reduction, drug cessation [dose Breakdown of changes

delay], discontinuation]

Stratification Outcome [Recovered/resolved,

item 2 : : recovering/resolving, not

recovered/not resolved,

recovered/resolved with sequelae,

fatal, unknown]

[Absent, present]

Total

The subjects in the above analysis will be stratified with Stratification Item 1 (this Method of

Analysis: product), and the frequency of the number of adverse drug reactions/infections will

be tabulated for each stratum in Stratification Item 2.

The same tabulation will be performed for AVD (Doxorubicin hydrochloride,

Property of Fakeda. For non-co vinblastine sulfate, and dacarbazine).

### 6 Efficacy analysis

### 6.1 Antitumor response after the end of frontline therapy

Analysis Patients in the efficacy analysis population for whom antitumor response was

population: assessed

Analysis item: Antitumor effect [With PET assessment, without PET

assessment, total]

Method of For each of the above analysis items, frequency of assessment results will be

Analysis: tabulated for patients in the efficacy evaluation set for whom antitumor response

has been assessed to calculate the response rate. In addition, a band graph will be prepared for the above analysis results. This tabulation will be performed for the entire population and patients excluding those who received a dose exceeding the

approved dose.

## 6.2 Antitumor effect after the end of frontline therapy by patient background factor and treatment factor

Analysis Patients in the efficacy analysis set for whom antitumor response was assessed

population:

Analysis item: Antitumor effect [With PET assessment, without PET

assessment, total]

Stratification Sex [Male, female]

item:

Property of Lakedai. Fc

Age (years)  $[Min \le -18, 18 \le -30, 30 \le -18]$ 

< 40, 40 <= - < 50, 50 <= - < 60, 60

<= - < 70, 70 <= - < 80, 80 <= - <=

Max]

Time from diagnosis of Hodgkin's [From the current month, the following

lymphoma to first dose of Adcetris month, and the second and subsequent

(months) months]

Lesion site (multiple counting) [Lymph nodes, spleen, liver,

lung,bone,central nervous system,

bone marrow, skin, others]

Clinical Stage (Ann Arbor [Stage I, II, III, IV, unknown]

Classification)

Presence or absence of B symptoms [Absent, present]

ECOG Performance Status [0, 1, 2, 3, 4]

Treatment classification (at the start of [Outpatient/inpatient]

treatment with Adcetris)

Presence or absence of complications [Absent, present] Presence or absence of concomitant [Absent, present] [Min <= - < 40.0, 40.0 <= - < 50.0, 50.0 <= - < 60.0, 60.0 <= - < 70.0 <= - <= Max \*\*

[M: renal impairment Presence or absence of concomitant [Absent, present] hepatic impairment Presence or absence of medical history [Absent, present, unknown] Body weight (kg)  $Min \le - < 18.5, 18.5 \le - < 25.0,$ BMI  $(kg/m^2)$ 25.0 <= - < 30.0, 30.0 <= - <= [Min <= - < 0.6, 0.6 <= - < 0.9, 0.9 Adcetris initial dose (mg/kg) Adcetris dose of mean (mg/kg) administration Adcetris dose (mg/kg/2weeks) Presence or absence of early G-CSF [Absent, present] administration

Method of Analysis:

For each of the above analysis items, the frequency of assessment results will be tabulated by stratum of the stratification items for patients who have been assessed for antitumor effect among the patients evaluable for efficacy, and the onse rate population and approved dose. response rate will be calculated. This tabulation will be performed for the entire population and patients excluding those who received a dose exceeding the

### Adverse reactions and infections in the additional pharmacovigilance plan

### Adverse reactions and infections included under the additional pharmacovigilance plan (Attached Form 12)

Analysis Safety analysis population

population:

Analysis item: Adverse reactions corresponding to safety specifications (important identified

risks)

Stratification [Serious, non-serious] Seriousness

item:

For the above analytical variable, the following analyses should be performed for Analytical

method: each of the subgroups of the stratification factors, in accordance with (Note) 1~4

of Form 12 in the Attachment of PSEHB/PED Notification No. 0325 No. 10

dated March 25, 2020.

(1) Number of subjects with events and the incidence of them

Property of Takeda. For non-commercial use only and The order of description of the risk name and risk name shall be in accordance

with the definition described in Important Identified Risks.

### Case summary in post-marketing surveillance

# act to the applicable reims of Use applicable reims of Use Case summary in post-marketing surveillance (Attached form 16)

Subjects to be CRF collected cases

analyzed:

Analysis item: Case No.

Name of medical institution

Sex

Age

Reason for use (Disease code, disease name)

Concomitant conditions (Disease code, disease name)

Route of administration

Maximum dose

Mean dose

Unit

Duration of use (duration of treatment with Adcetris)

Concomitant medicinal products (Drug Code, Drug Name)

Degree of effect

Adverse Reactions (Disease code, disease name, and outcome)

CRF number

withdrawal

Reason for withdrawal

G-CSF Early administration of drug product

For the above analysis items, a list will be prepared in accordance with the Analytical

Guidelines for Preparation of the Reexamination Data Entry File issued by method: Property of Fakeda. For not

PSEHB/PED Notification No. 1119 No. 3 dated November 19, 2020.

| version | date | Author/reviewer | comment |
|---------|------------|-----------------|----------------------------------|
| Version | 2023.01.26 | | Preparation of the first version |

Properly of Takeda: For non-commercial use only and subject to the applicable Temps of Use

LORO Eye

Dose

Inspection

Name

Sponsor

Property of T

mercial use only and subject to the applicable Tarms of Use

Original:

Prepared on September 7, 2023

### TABLE OF CONTENTS

| 1 Definition of Terms, etc | .2 |
|---|---|
| 1.1 List of Terms and Abbreviations | 2 |
| 1.2 Populations for Analyses | .4 |
| 1.3 digits to be displayed | 5 |
| 1.4 Important identified risks, important potential risks, and important missing information | 6 |
| (2) Patient characteristics | .7 |
| 2.1 Patient characteristics by early use or prophylactic use of G-CSF preparations | ~ > |
| (3) Matters related to safety | |
| 3.1 Data on adverse drug reactions/infections | <b>( 0</b> |
| 3.1.1 Occurrence Status of Adverse Reactions • Infections by the Presence or Absence of Early Administration or Prophylactic Administration of G-CSF Preparations (This | |
| Adverse reactions, etc. that occurred within 14 days after the start of administration of the drug) | .8 |
| 3.2 Occurrence Status of Adverse Reactions/Infections by Patient Background and Treatment Factor | .9 |
| 3.2. 1 Occurrence Status of Adverse Reactions • Infections by Patient Background Factor and Treatment Factor (Start of this drug Treatment) | |
| Adverse reactions, etc. that occurred within 14 days after the start of study treatment | .9 |
| 3.22 Occurrence Status of Adverse Reactions • Infections by Sex (Adverse Reactions that Occurred within 14 Days after the Start of the | nis |
| drug Treatment) | |
| Use, etc.) | 10 |
| 3.2. (3) Occurrence of ADRs • Infections by age group (Occurred within 14 days after the start of this drug treatment) ADVERSE REACTIONS, etc1 | 1 |
| 3.2, 4 Occurrence status of ADRs • Infections by presence or absence of concurrent renal impairment (14 days after the start of this drug treatment) | |
| Adverse reactions, etc. that occurred by the time of onset)1 | 1 |
| 3.2.5 Occurrence Status of ADRs • Infections by Presence or Absence of Concurrent Hepatic Impairment (14 days after the start of the drug treatment) | is |
| Adverse reactions, etc. that occurred by the time of onset) | 11 |
| 3.3 Occurrence Status of ADRs • Infections by Seriousness, CTCAE Grade (Worst Value), and Outcome (Administration of this drug | |
| Adverse reactions, etc. that occurred by 14 days after the start of administration) | |
| [4] Re-output of the final analysis figures/tables (replacement) | 13 |
| 4.1 Patient characteristics | 13 |
| 4.2 Occurrence Status of Adverse Drug Reactions/Infections by Patient Background Factor and Treatment Factor | |
| 4.3 Antitumor effect after the end of frontline therapy by patient demographics and treatment factors1 | 5 |
| Preparation history (version control) | 17 |
| Property of Takeda: For non-com. | |
| Operty of Tro | |

### 1 Definition of Terms, etc.

### 1.1 List of Terms and Abbreviations

- •this drug: Adcetris for Intravenous Drip Infusion 50 mg is abbreviated as this drug.
- •Adverse Event: AE occurred after administration of this drug.
- •Adverse reactions, etc.: An abbreviation of the term "adverse reactions infections." Adverse events that are not "not related" to this drug as
- The Important Medical Events List is used as the Medically Significant AE List, and events listed in the MedDRA code list (PT code) are handled as serious even if the investigator's assessment is "non-serious."

  Not related to this drug: An AE that is not related to this drug.

  Mot related to this drug: An AE that is not related. •Serious adverse events: Adverse events assessed as "serious" by the investigator. Takeda

- •Summary statistics: A collective term for sample size, mean, standard deviation, maximum, minimum, and quartiles.

  •Patients whose CRFs were not collected: Registered patients whose CRFs were not collected.

  •Patients whose CRFs were collected: Registered patients whose CRFs were collected.

  •Days after administration: Day -1 :- '
  drug to • Days after administration: Day -1 is defined as the day before the start date of this drug treatment and Day 1 is defined as the start date of this drug treatment.
- •Duration of treatment with this drug (days): end date of treatment with this drug (day): start date of treatment with this drug +1
- •Timing of onset of an adverse event (or adverse drug reaction, etc.): The date of onset of the adverse event (or adverse drug reaction, etc.) will be calculated as the start date of the first administration of one drug +1.
- •Time from Hodgkin's lymphoma diagnosis to first dose of this drug:
  - •Actual number (months) = (Year of the first administration of this drug Year of the diagnosis of Hodgkin's lymphoma) X12+ (Month of the first administration of this drug - Month of the diagnosis of Hodgkin's lymphoma) If the month of the diagnosis is unknown, January of the year will be used for calculation.
- Patients complicated with renal impairment: Takeda MedDRA query (Hereinafter referred to as TMQ) in the field of disease name

Complications applicable to "Disease" are listed.

- •Patients complicated with hepatic impairment: Patients in whom a complication corresponding to MedDRA standard query (Hereinafter referred to as SMQ) code 20000005 (liver disorder SMQ [scope: narrow]) is entered in the disease name field.
- Property of Fakedai. BMI (kg/m  $^{2}$ ): Calculated as weight (kg)/height (m)  $^{2}$  (rounded to the first decimal place).

- Early dose: G-CSF is administered within 5 days of the first dose of this drug.
- Non-early dose: G-CSF is administered on or after Day 6 of the first dose of this drug.
- Administration of a G-CSF preparation was administration.

  Administration of the start of this drug and have not included in the prophylactic administration.

  Administration other than prophylactic administration: The first dose of G-CSF preparation was administration was administration or after the onset of an AE.

  No prophylactic administration: Patients without G-CSF preparation and patients receiving only nor this drug administration: Day 1 of starting this drug +1 However, G-CSF.

- Properly of Takeda. For noncommercial use only and subject to the property of Takeda. this drug +1 However, G-CSF preparations should be administered from the first dose of this drug to before the second dose.

### 1.2 Populations for Analyses

As the analysis population of the general drug use-results survey, the "subjects for safety evaluation" and the "subjects for efficacy evaluation" will be defined. This analysis set will be defined as follows:.

property of Takeda. For noncommercial use only and subject to the property of takeda.

Property of Takeda. For non-commercial use only and subject to the applicable Temes of Use

5
- Properly of Lakeder, for non-confiner cial use only and subject to the applicable Latines of Use

6

## (2) Patient characteristics

## 2.1 Patient characteristics by early use or prophylactic use of G-CSF preparations

Analysis population: Subjects evaluable for safety

Analysis item: Sex

Age (years)

[Male, female]

[Min <=- < 18,18 <= - < 30, 30 <=-< 40, 40 <= - <

50, 50 <= - < 60, 60 <= - < 70, 70 <= - < 80, 80

<=- <=Max]

[Min <= - < 65, 65 <= - <= Max][From the

current month, the following month, and the

month after next]

Time from diagnosis of Hodgkin's lymphoma

to first dose of this drug (months)

Disease site (multiple counting)

[Lymph nodes, spleen, liver, lung, bone, CNS,

bone marrow, skin, others]

[Oral stage, stage B, stage B unknown]

[Absent, present]

[0,1,2, 3, 4]

[Outpatient/inpatient]

Absent, Present] Absent, Present] Absent,

Present] Absent]

[Absent, present, unknown]

[Min <= - < 40.0, 40.0 <= - < 50.0,50.0 <= - < 60.0,

60.0<= - < 70.0,70.0 <= - <= Max, not

measured]

[Min <=- < 18.5, 18.5 <= - < 25.0,25.0 <= - < 30.0,

30.0 <=- <= Max

Absent, Present]

Absent, Present] Absent, Present] Absent,

Present] Absent]

Clinical stage (Ann Arbor staging) Presence or absence of B symptoms

**ECOG Performance Status** 

Treatment category (at the start of this drug

treatment) Complications

Presence or absence of concurrent renal

impairment

Presence or absence of concurrent hepatic

impairment

Presence or absence of medical history

Weight (kg)

BMI(kg/m2) Breastfeeding status (females only)

Presence or absence of early administration of

G-CSF preparations

Presence or absence of prophylactic administration of G-CSF preparations

For the above analytical variables, in each of the subgroups of stratification factors (early administration of G-CSF preparations

Frequency tabulation of discrete data and summary statistics of continuous data will be calculated by the presence or absence of and the presence or absence of prophylactic administration of G-CSF preparations.

7

## (3) Matters related to safety

### 3.1 Occurrence status of adverse reactions/infections

3.1.1 Occurrence Status of Adverse Reactions • Infections by Presence or Absence of Early Administration or Prophylactic Presence of early administration of G-CSF preparations [Absent, present]
Presence or absence of prophylactic administration of G-CSF preparations [Absent, present]
The above analysis items were analyzed by the presence or absence of early administration of G-CSF preparations.
The following analyses will be performed by the presence or absence of prophylactic administration of the drug product.

(1) Number of patients with adverse administration of G-CSF preparations. Administration of G-CSF Preparations (e.g., Adverse Reactions that Occurred within 14 Days after the Start of this drug Treatment)

Analysis population:

Analysis item:

Analytical method:

Stratification item:

and by the presence or absence of early administration of G-CSF preparations.

- administration of this drug
- (2) Number of adverse drug reactions, etc. that occurred by 14 days after the start of administration of this
- (3) Incidence of adverse drug reactions, etc. that occurred within 14 days after the start of administration of this drug
- (4)  $Types\ of\ adverse\ drug\ reactions,\ etc.\ that\ occurred\ within\ 14\ days\ after\ the\ start\ of\ administration\ of\ this$

The calculation method for each analysis is as follows [Number of patients with adverse reactions, etc.]

- Number of patients with adverse reactions, etc. [Number of adverse reactions]
- Number of adverse drug reactions, etc. that occurred. If the same adverse drug reaction, etc. occurred multiple times in the same patient, the total number of events will be tabulated.

[Incidence of adverse reactions, etc.]

- Calculate with the number of patients with adverse drug reactions/number of patients evaluated for safety X100. [Types of adverse reactions]
- Adverse drug reactions will be coded using MedDRA/J. It will be roughly classified by SOC and tabulated by PT. SOC of "investigations" will be summarized by HLGT (Sort in ascending order of HLGT code, but do not output) and PT.
- In SOC, the number of patients with adverse drug reactions, etc. and the incidence will be described in SOC internationally agreed order. A subject with multiple occurrences of an event within an SOC should be counted only once for that SOC.
- Property of Takedai. For not By PT, the number of patients with adverse drug reactions, etc. and the incidence will be described in ascending order of PT codes. A subject who experienced the same PT more than once should be counted as 1 subject with the PT.

## 3.2 Occurrence Status of Adverse Reactions/Infections by Patient Background and Treatment Factor

# 3.2. 1 Occurrence of adverse drug reactions/infections by patient background factor and treatment factor (e.g., adverse drug reactions [Min <=- < 18,18 <= - < 30, 30 <= 6, 50 <= - < 60, 60 <= - < 76 = Max] that occurred within 14 days after the start of administration of this drug)

Analysis population:

Subjects evaluable for safety

Analysis item:

Adverse reactions, etc. that occurred within 14 days after the start of administration of this drug

Stratification item: Sex

[Male, female]

Age (years)

< 40, 40 <= - < 50, 50 <= - < 60, 60 <= - < 70, 70

<= - < 80, 80 <=- <=Max]

[Min <= - < 65, 65 <= - <= Max][From the]current month, the following month, and the

month after next]

Time from diagnosis of Hodgkin's lymphoma

to first dose of this drug (months) Disease site (multiple counting)

Clinical stage (Ann Arbor staging) Presence or absence of B symptoms

**ECOG Performance Status** 

Treatment category (at the start of this drug

treatment) Complications

Presence or absence of concurrent renal

impairment

Presence or absence of concurrent hepatic

impairment

Presence or absence of medical history

Weight (kg)

[Lymph nodes, spleen, liver, lung, bone, CNS,

bone marrow, skin, others]

[Oral stage, stage B, stage B, stage B unknown]

[Absent, present] [0,1,2,3,4]

[Outpatient/inpatient] [Absent, present]

[Absent, present]

Absent, Present]

Absent, present, unknown]

[Min <= - < 40.0, 40.0 <= - < 50.0, 50.0 <= - < 60.0,

60.0<= - < 70.0,70.0 <= - <= Max, not measured]

[Min <=- < 18.5, 18.5 <= - < 25.0,25.0 <= - < 30.0,

30.0 <=- <= Max

[Min <= - < 0.6, 0.6 <= - < 0.9, 0.9 <=

- < 1.2, 1.2,1.2 < - <= Max]

[Min <= - < 0.6, 0.6 <= - < 0.9, 0.9 <=

- < 1.2, 1.2,1.2 < - <= Max]

[Min <= - < 0.6, 0.6 <= - < 0.9, 0.9 <=

- < 1.2, 1.2,1.2 < - <= Max]

Absent, Present]

This drug loading dose (mg/kg)

Mean dose of this drug per administration (mg/kg)

Property of Fakeda. For hox This drug dose per 2 weeks (mg/kg/2 weeks) Presence or absence of early administration of G-CSF

preparations

Analytical method:

For the above analytical variable, the following analyses should be performed for each stratum of the stratification factor.

 $Number of patients with adverse drug \ reactions, etc. \ that occurred by 14 \ days \ after \ the \ start \ of \ administration \$ 

Incidence of adverse drug reactions, etc. that occurred by 14 days after the start of administration of this drug The \* ems of Use method of counting in each analysis is as follows.

[Number of patients with adverse reactions, etc.]

Number of patients with adverse reactions, etc. [Incidence of adverse reactions, etc.] Calculate with the number of patients with adverse drug reactions/number of patients evaluated for safety X100.

## 3.2. 2 Occurrence status of ADRs • Infections by sex (ADRs that occurred within 14 days after the start of administration of this drug, etc.)

Analysis population:

Subjects evaluable for safety

Analysis item:

Adverse reactions, etc. that occurred within 14 days after the start of administration of this drug

[Male, female]

Stratification item: Sex Analytical method: stratification factor.

For the above analysis set, the following analyses will be performed for each stratum of the

 $Number of patients with adverse drug \ reactions, etc. \ that occurred \ by \ 14 \ days \ after \ the \ start \ of \ administration \ of \ administratio$ this drug

Number of adverse drug reactions, etc. that occurred by 14 days after the start of administration of this drug Incidence of adverse drug reactions, etc. that occurred within 14 days after the start of administration of this drug Type of adverse drug reactions, etc. that occurred by 14 days after the start of administration of this drug The method of counting in each analysis is as follows.

[Number of patients with adverse reactions, etc.]

- Number of patients with adverse reactions, etc. [Number of adverse reactions]
- Number of adverse drug reactions, etc. that occurred. If the same adverse drug reaction, etc. occurred multiple times in the same patient, the total number of events will be tabulated.

[Incidence of adverse reactions, etc.]

- Calculate with the number of patients with adverse drug reactions/number of patients evaluated for safety X100. [Types of adverse reactions, etc.]
- Adverse drug reactions will be coded using MedDRA/J. It will be roughly classified by SOC and tabulated by PT. SOC of "investigations" will be summarized by HLGT (Sort in ascending order of HLGT code, but do not
- In SOC, the number of patients with adverse drug reactions, etc. and the incidence will be described in SOC internationally agreed order. A subject with multiple occurrences of an event within an SOC should be counted only once for that SOC.

Property of akedai. By PT, the number of patients with adverse drug reactions, etc. and the incidence will be described in ascending order of PT codes. A subject who experienced the same PT more than once should be counted as 1 subject with the

# 323 Onset status of ADRs • infections by age group (ADRs, etc. that occurred within 14 days after the start of administration of this

Analysis population: Subjects evaluable for safety

Adverse reactions, etc. that occurred within 14 days after the start of administration of this drug Analysis item:

[Min <=- < 18,18 <= - < 30, 30 <=-Stratification item: Age (years) < 40, 40 <= - < 50, 50 <= - < 60, 60

<=-< 70, 70 <= - < 80, 80 <=- <=Max]

[Min <= - < 65, 65 <= - <= Max]

applicable rems of Use Analytical method: For the above analytical variable, the same analyses as those described in Section 3.2.2 were performed for each

stratum of the stratification factor.

Perform.

## 3.2. 4 Incidence of ADRs • Infections by presence or absence of concurrent renal impairment (ADRs, etc. that occurred within 14 days after the start of administration of this drug)

Subjects evaluable for safety Analysis population:

Adverse reactions, etc. that occurred within 14 days after the start of administration of this drug Analysis item:

[Absent, present] Stratification item: Presence or absence of concurrent renal impairment

For the above analysis set, the same analyses as those described in Section 3.2.2 were performed for each stratum of the same analysis set in the same analysis set in the same analysis are the same analysis as those described in Section 3.2.2 were performed for each stratum of the same analysis set, the same analysis are those described in Section 3.2.2 were performed for each stratum of the same analysis are those described in Section 3.2.2 were performed for each stratum of the same analysis are tAnalytical method: only and

the stratification factor

Perform.

## 3. 2.5 Occurrence status of ADRs • Infections by presence or absence of concurrent hepatic impairment (ADRs, etc. that occurred within 14 days after the start of administration of this drug)

Subjects evaluable for safety Analysis population:

Analysis item: Adverse reactions, etc. that occurred within 14 days after the start of administration of this drug

Stratification item: Presence or absence of concurrent hepatic impairment [Absent, present]

Perform.

Perform. For the above analysis set, the same analyses as those described in Section 3.2.2 were performed for each stratum of

3.3 Occurrence Status of Adverse Reactions • Infections by Seriousness, CTCAE Grade (Worst Value), and Outcome (Adverse Reactions, etc. that Occurred within 14 Days after the Start of this drug Treatment) Analysis Set: Subjects evaluable for safety

Analysis item: Adverse reactions, etc. that occurred within 14 days after the start of administration of this drug

Stratification item: Total

Seriousness [Serious, non-serious] CTCAE Grade (worst value) [Grade3, Grade4, Grade5]

Outcome [recovered/resolved, recovering/resolving, not

recovered/not resolved, recovered/resolved but later]

ermsofuse Presence of residual disease, death (due to this event),

In the above analysis

unknown] Analysis method:

population, subjects with or without early administration of G-CSF preparations and subjects with G-CSF

For each of the stratification factors with or without prophylactic administration of the product, the same analyses as those in Section 3.1.1 will be performed. A subject who experienced the same SOC/PT more than once should be counted as 1 subject in the SOC/PT. However, 1 subject within the same SOC will be included in the study according to the following order of priority, and 1 subject within the same PT will be included in the study according to the following order of priority for any of the stratification factors.

Seriousness: Serious - Non-serious

Property of Takeda. For noncommercial use only and subject of takeda. Outcome: Death (due to this event) Recovered once with sequelae 1 Not recovered/Not resolved T Recovering/Resolving T Unknown

12

## [4] Re-output of the final analysis figures/tables (replacement)

## 4.1 Patient characteristics

Analysis population: Subjects evaluable for safety

Analysis item: Sex

[Male, female] Age (years)

[Min <=- < 18,18 <= - < 30, 30 <=-< 40, 40 <= - < 50, 50 <= - < 60, 60 <=-< 70, 70 <= - < 80, 80 <=- <=Max]

[From the current month, the following month?

and the month after next]

Time from diagnosis of Hodgkin's lymphoma

to first dose of this drug (months) Disease site (multiple counting)

[Lymph nodes, spleen, liver, lung, bone, CNS, bone marrow, skin, others]

[Oral stage, stage B, stage B unknown]

[Absent, present]

[0,1,2,3,4]

Clinical stage (Ann Arbor staging) Presence or absence of B symptoms

**ECOG Performance Status** 

[Outpatient/inpatient] [Absent, present]

[Absent, present] [Absent, present]

Treatment category (at the start of this drug

treatment) Complications

Absent, present, unknown] Presence or absence of concurrent renal

impairment

Presence or absence of concurrent hepatic

[Min <=- < 18.5, 18.5 <= - < 25.0,25.0 <= - < 30.0,

Presence or absence of medical history

Min <= - < 40.0, 40.0 <= - < 50.0,50.0 <= - < 60.0,

 $60.0 \le - < 70.0, 70.0 \le - \le Max, \text{ not measured}$ 

30.0 <=- <= Max

Absent, Present] Breastfeeding status (females Absent, Present]

pnly) For the above analytical variables, frequency tabulation of discrete data and continuous data

Summary statistics will be calculated.

4.2 Occurrence Status of Adverse Drug Reactions/Infections by Patient Background Factor and Treatment Factor

Analysis population: Subjects evaluable for safety

Analysis item: Adverse reactions, etc.

Stratification item: \$\doc{\forall}{g} ex [Male, female]

> [Min <=- < 18,18 <= - < 30, 30 <=-Age (years)

> > < 40, 40 <= - < 50, 50 <= - < 60, 60

<=-< 70, 70 <= - < 80, 80 <=- <=Max]

[From the current month, the following month, and the month after next]

Time from diagnosis of Hodgkin's lymphoma to first dose of this drug (months)

Disease site (multiple counting)

icable Terms of Use [Lymph nodes, spleen, liver, lung, bone, CNS,

bone marrow, skin, others]

stage B, stage B, stage B, unknown

[Absent, present]

[0,1,2,3,4]

[Outpatient/inpatient]

Absent, Present]

Absent, Present]

Absent, Present]

[Absent, present, unknown]

[Min <= - < 40.0, 40.0 <= - < 50.0, 50.0 <= - < 60.0,

60.0<= - < 70.0,70.0 <= <= Max, not measured]

[Min <=- < 18.5, 18.5 <=- < 25.0,25. <= - < 30.0,

30. <= - <= Max

[Min <= < 0.6, 0.6 <= - < 0.9, 0.9 <=

- < 1.2, 1.2,1.2 < - <= Max]

Min <= - < 0.6, 0.6 <= - < 0.9, 0.9 <=

- < 1.2, 1.2,1.2 < - <= Max]

Min <= - < 0.6, 0.6 <= - < 0.9, 0.9 <=

- < 1.2, 1.2,1.2 < - <= Max]

Absent, Present]

Clinical stage (Ann Arbor staging)

Presence or absence of B symptoms

**ECOG Performance Status** 

Treatment category (at the start of this drug

treatment) Complications

Presence or absence of concurrent renal

impairment

Presence or absence of concurrent hepatic

impairment

Presence or absence of medical history

Weight (kg)

BMI(kg/m2)

This drug loading dose (mg/kg)

Mean dose of this drug per administration (mg/kg)

This drug dose per 2 weeks (mg/kg/2 weeks) Presence or absence of early administration of G-CSF

preparations

Analytical method:

For the above analytical variable, the following analyses should be performed for each stratum of the stratification factor.

Number of patients with adverse reactions, etc.

Incidence of adverse drug reactions

The calculation method for each analysis is as follows.

[Number of patients with adverse reactions, etc.]

•Number of patients with adverse reactions, etc.

[Incidence of adverse reactions, etc.]

 $Calculate\ with\ the\ number\ of\ patients\ with\ adverse\ drug\ reactions/number\ of\ patients\ evaluated\ for\ safety\ X100.$ 

## 4.3 Antitumor effect after the end of frontline therapy by patient demographics and treatment factors

Analysis population: Patients whose antitumor effect was assessed among the patients evaluated for efficacy

Analysis item: Antitumor effect

total]

[Male, female]

Stratification item: Sex

Age (years)

[Mln v=- < 18,18 v= - < 30, 30 v=

[With PET assessment, without PET assessment,

v= - v 70, 70 v= - v 80, 80 v= - v=

Max]

< 40, 40 v= - v 50, 50 v= - v 60, 60 , 80 v= - v=

nonth +' [From the current month, the following month, and the month after next]

Time from diagnosis of Hodgkin's lymphoma to first dose of this drug (months) Disease site (multiple counting)

[Lymph nodes, spleen, liver, lung, bone, CNS,

[Oral stage, stage B, stage B, stage B unknown]

Absent, Present]

Treatment category (at the start of this drug

treatment) Complications

Presence or absence of concurrent renal

Clinical stage (Ann Arbor staging)

**ECOG Performance Status** 

Presence or absence of B symptoms

impairment

Presence or absence of concurrent hepatic

impairment

Presence or absence of medical history

bone marrow, skin, others]

[0,1,2,3,4]

[Outpatient/inpatient]

Absent, Present] Absent, Present] Absent, Present]

[Absent, present, unknown] [Min v= - v 40.0, 40.0 v= - v 50.0,

50.0 v= - v 60.0, 60.0v= - v 70.0, 70.0 v= -v= Max, not measured

25. v = -v 30.0, 30. v = -v = Max

[Min v= -v 0.6, 0.6 v= -v 0.9, 0.9 v=-v 1.2,

[Min v= - v 18.5, 18.5 v= - v 25.0,

Mean dose of this drug per administration (mg/kg)

Min v= - v 0.6, 0.6 v= - v 0.9, 0.9 v= -v 1.2, 1.2,1.2 v - v= Max]

1.2,1.2 v - v = Max

Min v= - v 0.6, 0.6 v= - v 0.9, 0.9 v=

-v 1.2, 1.2,1.2 v - v= Max]

Absent, Present]

Property of Takeda. For non-commercial This drug dose per 2 weeks (mg/kg/2 weeks) Presence or absence of early administration of G-CSF

For each of the above analysis items, the tumor response was assessed in the efficacy analysis set.

Frequency tabulation of assessment results by stratum of stratification items in patients who were assessed

will be performed to calculate the response rate. This tabulation will be performed for the overall population and the

Properly of Takeda. For non-confine cial use only and subject to the applicable Tames of Use

## Preparation history (version control)

| Version | Date | Author/Reporter | Comments |
|---|---|---|---|
| | | | Preparation of initial version |
| Original<br>Version | 2023.9.7 | | [4] Regarding the re-output (replacement) of the final analysis figures and tables, there was an error in the derivation method for the "period category from the diagnosis of Hodgkin's lymphoma to the first dose of this drug" at the final analysis. Therefore, correction of the derivation method and reoutput of related figures and tables were planned. |

A med

- a med

- a m